CLINICAL TRIAL: NCT04454593
Title: Novel Method for Diagnosing Lateral Patellar Compression Syndrome Using X-ray: a Retrospective Case-Control Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019464
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Lateral Patellar Compression Syndrome
Keywords: Lateral patellar compression syndrome; Lateral patellar curvature angle; Patellar axial radiographs; The area under the curve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lateral patellar compression syndrome: Patients diagnosed with lateral patellar compression syndrome between February 2016 and April 2019
  Interventions: Other: no intervention
- patellar dislocation: Patients diagnosed with patellar dislocation between February 2016 and April 2019
  Interventions: Other: no intervention
- meniscus tear: Patients diagnosed with meniscus tear between February 2016 and April 2019
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study,with no intervention

SUMMARY:
This study evaluates whether the patellar axial radiograph of lateral patellar curvature angle （LPCA）with knee flexion at 30 ° can be used as a new diagnostic surrogate of lateral patellar compression syndrome（LPCS）. We believe that the new index LPCA has high sensitivity and specificity in initial diagnosis of LPCS using axial patellar radiograph with knee flexion at 30 ° , and has high application value.

DETAILED DESCRIPTION:
Background: A well-established reference is lacking for diagnosing lateral patellar compression syndrome (LPCS), and this diagnosis currently depends on clinicians' subjective judgment and several examination results. X-rays are primarily used to diagnose LPCS, but they have low detection rates of patellar tilt using the congruence angle (CA) and patellar tilting angle (PTA).

Purpose: To investigate whether patellar axial radiography of the lateral patellar curvature angle (LPCA) of knee in 30° flexion can diagnose LPCS.

Methods: We enrolled 87 patients between 2016 and 2019 and divided them as per diagnosis into three groups of 29 each: LPCS, patellar dislocation (PD, control), and meniscus tear (MT, negative control) groups. A senior radiologist and the chief physician of sports medicine examined their patellar axial radiographs of the knee in 30° flexion using a computer imaging system, measuring LPCA, PTA, and CA. Univariate analysis of variance and Kruskal-Wallis H test were used to compare measurement data with normal distribution and non-normal distribution, respectively. Bonferroni correction was used to analyze different indicators for different groups. The area under the curve (AUC) was calculated to verify the value of LPCA in initial diagnosis of LPCS.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as LPCS ，MT and PD respectively

Exclusion Criteria:

* patients with ligament injury, malunion of patella fracture, free bodies in the joint, surgical contraindications, and with both knees affected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We enrolled 87 patients between 2016 and 2019 and divided them as per diagnosis into three groups of 29 each: LPCS, patellar dislocation (PD, control), and meniscus tear (MT, negative control) groups.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
lateral patellar curvature angle | between 2016 and 2019
  lateral patellar curvature angle in three groups was compared

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yu-ping, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No